CLINICAL TRIAL: NCT02526706
Title: VisionBlue for the Assessment of Filtering Bleb Functioning During Cataract Surgery
Brief Title: Using a Type of Blue Dye to Observe Bleb Function During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Marlene Moster, MD, MD, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15-494
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Bleb filtration; VisionBlue
MeSH Terms: conditions — Glaucoma | interventions — Trypan Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glaucoma Study Group (Experimental): Glaucoma patients scheduled for trabeculectomy were recruited for this study and VisionBlue dye is injected prior to the surgery.
  Interventions: Other: VisionBlue

INTERVENTIONS:
Other: VisionBlue — VisionBlue is a staining solution designed to assist in making complete capsulorhexis during cataract surgery. The dye is injected into the anterior chamber via a paracentesis port and stains the anterior lens capsule, assisting in adequate visualization of the anterior lens capsule. This study proposes to explore the use of VisionBlue during cataract surgery as a means to assess functioning of an existing filtering bleb placed during prior trabeculectomy in patients with glaucoma.

SUMMARY:
The investigators aim to conduct a prospective clinical pilot study to investigate the use of VisionBlue staining administered during cataract surgery to 20 patients with history of trabeculectomy for glaucoma as a means to assess functioning of an existing filtering bleb. The investigators also aim to develop a standard classification system for assessing filtering bleb function during cataract surgery.

DETAILED DESCRIPTION:
Twenty (20) patients with history of trabeculectomy who have been scheduled for cataract extraction with posterior chamber intraocular lens implant, will be recruited from Wills Eye Hospital Glaucoma Service.

Subjects will undergo a comprehensive ophthalmic evaluation prior to scheduling cataract surgery. The following data will be recorded: Demographic information including age, race, and gender, Best corrected visual acuity, IOP measured by Goldmann applanation tonometry, Bleb morphology evaluation using the Indiana Bleb Appearance Grading Scale (IBAGS), Filtering bleb photographs and anterior segment OCT of the bleb will be taken at the baseline examination.

The patient will be taken to the operating room and will be prepped.Non-preserved Lidocaine (1%) will be injected into the anterior chamber for anesthesia, followed by injection of one complete vial of VisionBlue (0.5 mL). An injection of BSS will be administered through the paracentesis port until the IOP is approximately 20mHg (estimated by the surgeon by palpation), with a waiting period of 20 seconds. Another injection of BSS will then be administered to wash out the VisionBlue. A set of microscopic photographs will be taken through the intraoperative microscope following washout of VisionBlue, with bleb grading performed by the physician: 1+ to 4+ stain (based on standard set of photos).

Cataract extraction will then take place following typical phacoemulsification procedure. At the end of the case, after insertion of the intraocular lens implant into the capsular bag and removal of viscoelastic material from the eye, an additional set of microscope photographs will be taken and graded on same scale.

The time (in minutes) between the initial and the final bleb grading will be measured and recorded. Intraoperative complications will be recorded as well.

Follow-up of subjects will take place post-operatively at 1 day, 1 week, 1 month, 3 month, and 6 month follow-up visits. Color photos of bleb will be performed post-operatively at 1 day, 1 month, and 6 months. At each visit, we will also record the number of glaucoma medications, post-operative complications and need for re-operations.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients with history of previous trabeculectomy surgery who are scheduled for cataract surgery.
* Glaucoma defined as (both requirements must be met): 1) Characteristic glaucomatous disc damage as demonstrated by local narrowing, notching, or absence of the neuroretinal rim in the absence of disc pallor elsewhere. 2) Characteristic glaucomatous visual field (VF) deficits.
* Over 21 years of age

Exclusion Criteria:

* Intraocular surgery or laser procedure within 3 months prior to the planned cataract surgery.
* Active ocular infection or inflammation.
* History of glaucoma drainage device (tube-shunt) implantation.
* Allergy to VisionBlue or history of allergy to other ophthalmic dyes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) post surgery | 6 months
  IOP is measured pre and post operation and in all the follow up visits.
The Indiana Bleb Appearance Grading System (IBAGS) will be used for bleb grading | 6 months
  Evaluation based on pre-operative bleb photography will be compared to intraoperative VisionBlue bleb scoring by using Indiana Bleb Appearance Grading System (IBAGS) as a standard structured framework for comparison. The IBAGS method uses bleb photography to create a score based on bleb height (0 to 3), extent (0 to 3), vascularity (0 to 4), and Seidel test leakage (0 to 2).
Change in Glaucoma medication from pre to post surgery | 6 months
  Observe the changes in glaucoma medication after surgery procedure and at all follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Moster, MD, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Hospital, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No